CLINICAL TRIAL: NCT00367224
Title: Determining the Tolerance of Depigmented Skin to Targeted Phototherapy Using UVB in Patients With Vitiligo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Dermatologist, Henry Ford Health System
Other Study IDs: IRB3701
Record Dates: First submitted 2006-08-18; First posted 2006-08-22 (Estimated); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Vitiligo
Keywords: vitiligo; tolerance; ultraviolet B.
MeSH Terms: conditions — Vitiligo | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: 6 to 9 ultraviolet B treatments — Treatments with ultraviolet B with gradually progressive doses
  Other Names: phototherapy
Procedure: Skin biopsies — 4 mm punch biopsies of the skin
  Other Names: Skin biopsy, skin sample

SUMMARY:
The purpose of this study is to determine if vitiligo patients develop tolerance to ultraviolet light therapy, a type of treatment available for vitiligo.

DETAILED DESCRIPTION:
Patients with vitiligo received 6-9 ultraviolet B treatments, 2 to 3 times weekly. Minimal erythema dose (MED) testing was done at baseline and after all treatments; the percent change in MED was analysed as a measure of photoadaptation. The percent decrease in cyclobutane pyrimidine dimers (CPDs) over 24 hours after a single exposure of 1 MED was analysed on vitiliginous and normal skin.

ELIGIBILITY:
Inclusion Criteria:

For inclusion, the subject must:

1. Be at least 18 years old
2. Be otherwise healthy
3. Have a diagnosis of vitiligo affecting > 5% body surface area (BSA)
4. Have two depigmented lesions on opposite sides of the body that can be biopsied at the end of TARGETED UVB PHOTOTHERAPY treatment
5. Agree to abide by the Investigator's guidelines regarding photosensitizing drugs
6. Have a negative pregnancy test at baseline if female of childbearing potential
7. Be able to understand the requirements of the study, the risks involved, and is able to sign the informed consent form
8. Agree to follow and undergo all study-related procedures

Exclusion Criteria:

Subjects will be excluded if any of the following apply:

1. Women who are lactating, pregnant, or planning to become pregnant
2. Patients with a recent history of serious systemic disease
3. Patients with a known history of photosensitivity
4. Concomitant use of systemic or topical treatments for vitiligo. Patients must discontinue PUVA or oral corticosteroid therapy for 4 weeks prior to the start of any treatment. If a patient is taking any vitamins or dietary supplements, the patient must discontinue them for the duration of the study. Topical therapy such as corticosteroids, topical immunomodulators (e.g., Protopic or Elidel), vitamin D derivatives (e.g., Dovonex), or UVB phototherapy must be discontinued for 2 weeks prior to the start of study treatment.
5. Patients diagnosed to be immunosuppressed for any reason (e.g., HIV infection, lupus, cancer, organ transplant, or chronic use of oral immunosuppressive agents).
6. Any reason the investigator feels the patient should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat Hamzavi, Principal Investigator — Department of Dermatology, Henry Ford Health System
Locations (1):
- Department of Dermatology/Henry Ford Hospital, Detroit, Michigan, United States

REFERENCES:
- [Derived] Hexsel CL, Mahmoud BH, Mitchell D, Rivard J, Owen M, Strickland FM, Lim HW, Hamzavi I. A clinical trial and molecular study of photoadaptation in vitiligo. Br J Dermatol. 2009 Mar;160(3):534-9. doi: 10.1111/j.1365-2133.2008.08943.x. Epub 2008 Dec 5. PMID 19067714